CLINICAL TRIAL: NCT02173067
Title: Local Anesthesia With Epinephrine for Oral Surgery in Type 2 Diabetes Mellitus With Corornary Disease is Safe and Effective
Brief Title: Anesthesia With Epinephrine in Diabetes Patients is Safe and Effective
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: Odonto - Diabetes
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Disease
Keywords: Diabetes mellitus; Epinephrine; Anesthesia, Dental; lidocaine; Ambulatory Surgical Procedures
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: None Retained — Type 2 diabete mellitus (in use of insulin and/or hypoglicemic agents) with coronary disease adults patients who needes to have at least one posterior maxillary tooth extracted, according to oral examination and panoramic radiography.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2% lidocaine: 35 patients received 5.4 mL of 2% lidocaine.
- 2% lidocaine with epinephrine: 35 patients recieved 5.4 mL of 2% lidocaine with 1:100,000 epinephrine.

SUMMARY:
The purpose of this study is to investigate the variation in blood glucose levels, hemodynamic effects and patient anxiety score during tooth extraction in type 2 diabetes mellitus with coronary disease patient under local anesthesia with lidocaine 2% with and without epinephrine.

DETAILED DESCRIPTION:
This is a prospective randomized study including 70 diabetes with coronary disease patients that needed to be submitted to oral surgery. The study was double blind in relation to glycaemia measurements. Continuous monitoring of blood glucose levels for 24 hours was performed using the Minimed Continuous Monitoring System (CGMS, Medtronic). Patientes were randomized into two groups: 35 received 5.4 mL of 2% lidocaine and 35 received 5.4 mL of 2% lidocaine with 1:100,000 epinephrine. In addittion, hemodynamic effects (blood pressure and heart rate) and degree of anxiety were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes mellitus pharmacologically controlled (in use of insulin and/or hypoglycemic agents) Coronary disease -

Exclusion Criteria:

* Pregnant sepsis acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled pharmacologically controlled type 2 diabetes mellitus (in use of insulin and/or hypoglycemic agents) and with coronary disease adult patient who needed to have at least one posterior maxillary tooth to be extracted.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
varition in blood glucose levels during oral surgery with local anaesthesia (lidocaina and lidocaine with epinephrine) | 24 hours
  To asses the blood glucose levels the Continuous monitoring system (MiniMed CGMS, Medtronic) was employed. The MiniMed monitor was installed in the morning of the day before the surgery and the patient went to home. The patient returned to the hospital for the surgery 24 hours later and the monitor was retired one hour after the end of the oral surgery.

SECONDARY OUTCOMES:
Hemodynamic effects during the surgery with local anesthetia (lidocaine and lidocaine with epinephrine) | almost 3 hours
  Systolic blood pressure, diastolic blood pressur and heart rate were recorded by automatic sphygmomanometer (Microlife APA-P00001) in four times: one hour before the surgery, five minutes before the surgery, after anesthesia injection and one hour after the surgery.

OTHER OUTCOMES:
Anxiety levels during the oral surgery with local anesthesia (lidocaine and lidocaine and epinephrine) | almost 3 hours
  Anxiety levels was measurement by the Image Facial Scale at the times: one hour before the surgery, five minutes before the surgery and one hour after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela A Santos, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Unit of Dentistry, Heart Institute, São Paulo, São Paulo, Brazil